CLINICAL TRIAL: NCT04036201
Title: Minimum Effective Volume of Local Anesthetic for Peribulbar Block.Does it Differ With the Eyeball Axial Length?
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Walid Nofal, Assisstant Professor of Anesthesiology, Ain Shams University
Allocation: Non-Randomized | Model: Parallel | Masking: Double | Purpose: Health Services Research
Other Study IDs: FMASU R 41/2019
Record Dates: First submitted 2019-07-22; First posted 2019-07-29 (Actual); Last update posted 2019-10-22 (Actual); Status verified 2019-10

CONDITIONS: Peribulbar Block
Keywords: Peribulbar block; minimum effective volume; axial eye length
MeSH Terms: interventions — Bupivacaine; Hyaluronic Acid

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Group 1(22-24 mm) (Experimental): Group 1 (patients with axial length between 22 and 24 mm): received a mixture of bupivacaine 0.5% (3ml) + lidocaine 2% (3ml) + hyalurindase 150 IU (1 ml) to a total volume of 7 ml.
  Interventions: Drug: Bupivacaine
- Group 2(24.1-26 mm) (Experimental): Group 2 (patients with axial length between 24.1 and 26 mm): received a mixture of bupivacaine 0.5% (3ml) + lidocaine 2% (3ml) + hyaluronidase 150 IU (1 ml) to a total volume of 7 m
  Interventions: Drug: Bupivacaine

INTERVENTIONS:
Drug: Bupivacaine — peribulbar block
  Other Names: hyaluronic acid

SUMMARY:
The aim of this study is to calculate the minimum effective volume of local anesthetic for peribulbar block in patients undergoing cataract extraction surgery.

DETAILED DESCRIPTION:
The main goal of this study is to estimate the minimum effective volume(MEV90) of local anesthetic and hyaluronic acid given for local anesthesia of the eye for 2 different axial length groups of patients undergoing eye surgery. Volume assignment was carried out using a biased coin design (BCD) up-and-down sequential method (UDM), where the volume given to each patient depends on the response of the previous one. The MEV90 was calculated using isotonic regression with bias-corrected 95% confidence interval (CI) derived by boots trapping. The mean value of the estimate was obtained from 3000 bootstrap samples.

ELIGIBILITY:
Inclusion Criteria:

* we allocated adult patients aged 40-70 years, of both gender, American Society of Anesthesiologists (ASA) II - III, listed for elective cataract extraction using phaco emulsification technique with intraocular lens implantation surgery.

Exclusion Criteria:

* Patients known to have any systemic contraindications (as severe hypertension) or allergy to the local anesthetic, those who refused local anesthesia, high myopes (axial length > 26 mm), patients with a single eye, those with complicated vitreous hemorrhage, ocular infection, or associated glaucoma have been excluded.

Ages: 40 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 121 (Actual)
Dates: Start 2019-07-31 (Actual); Primary Completion 2019-10-10 (Actual); Study Completion 2019-10-10 (Actual)

PRIMARY OUTCOMES:
The minimum effective volume of local anesthetic of the eye in relation to the eyeball axial length. | 10 minutes
  The minimum effective volume of local anesthetic in peribulbar block in relation to the eyeball axial length.The minimum volume which will achieve adequate sensory and motor block within 10 minutes.

CONTACTS AND LOCATIONS:
Overall Officials: WALID Nofal, MD, Principal Investigator — Faculty of Medicine, Ain Shams University; Sanaa el Fawal, MD, Principal Investigator — Faculty of Medicine, Ain Shams University; Wail Abdelaal, MD, Principal Investigator — Faculty of Medicine, Ain Shams University; Eman Sabek, MD, Principal Investigator — National Centre of Radiation Research and Technology, Atomic Energy Authority
Locations (1):
- Faculty of Medicine ,Ain Shams University, Cairo, Cairo Governorate, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] El Fawal SM, Nofal WH, Sabek EAS, Abdelaal WA. Minimum effective volume of local anesthetic in peribulbar block: does it differ with the eyeball axial length? Braz J Anesthesiol. 2021 Nov-Dec;71(6):635-641. doi: 10.1016/j.bjane.2021.09.001. Epub 2021 Sep 22. PMID 34562489